CLINICAL TRIAL: NCT05915676
Title: Frequency Assessment of Leukocyte Immunoglobulin-like Receptors A3 In Ankylosing Spondylitis And Axial Psoriatic Arthritis Patients
Brief Title: Role of LILRA3 in Ankylosing Spondylitis and Axial Psoriatic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Adel Abdelmoez, Frequency Assessment of Leukocyte Immunoglobulin-like receptors A3 In Ankylosing Spondylitis And Axial Psoriatic Arthritis Patients, Assiut University
Other Study IDs: LILRA3 in AS, Axial psoriasis
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Leukocyte Immunoglobulin-like receptors A3 — Leucocyte immunoglobulin-like receptor A3 (LILRA3) belongs to a family of leucocyte receptors produced as a soluble molecule by monocytes and macrophages. (3) The function of LILRA3 remains obscure, but LILRA3 could bind to HLA class I molecules HLA-G and HLA- C (4) and may act as an antagonist on other LILRs or a soluble ligand to other receptors(5) Growing evidence shows that (LILRA3) is associated with many autoimmune disorders.(6) (7) The functional LILRA3 is a susceptibility factor for AS and axial psoriatic arthritis (axPsA) has not been investigated.

SUMMARY:
1. To evaluate the frequency of LILRA3 in Ankylosing spondylitis and Axial psoriatic arthritis patients.
2. To investigate the association of LILRA3 with Ankylosing spondylitis and Axial psoriatic arthritis disease activity and severity.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) is a complex inflammatory condition that affects the axial skeleton including the sacroiliac joints and the spine (1). It also affects peripheral joints and can be associated with extra-musculoskeletal manifestations including uveitis, psoriasis, and inflammatory bowel disease (1).

Axial spondyloarthritis include ankylosing spondylitis (AS), certain forms of psoriatic arthritis (PsA), reactive arthritis with axial involvement, and arthritis associated with inflammatory bowel disease (2).

The diagnosis of axSpA remains very challenging with years of delays attributed to several different factors. There is also a strong need to identify new serological biomarkers that can aid clinicians for diagnosis of axSpA.

Leucocyte immunoglobulin-like receptor A3 (LILRA3) belongs to a family of leucocyte receptors produced as a soluble molecule by monocytes and macrophages. (3) The function of LILRA3 remains obscure, but LILRA3 could bind to HLA class I molecules HLA-G and HLA- C (4) and may act as an antagonist on other LILRs or a soluble ligand to other receptors(5) Growing evidence shows that (LILRA3) is associated with many autoimmune disorders.(6) (7) The functional LILRA3 is a susceptibility factor for AS and axial psoriatic arthritis (axPsA) has not been investigated.

ELIGIBILITY:
Inclusion Criteria:Adult AS and axPsA patients <18 years Who fulfilled the Assessment of SpondyloArthritis international Society (ASAS) criteria for axSpA.

-

Exclusion Criteria:1-patients less than 18 years old

2-Individuals with other autoimmune diseases

-

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
LILRA3 in AS and Axial psoriatic arthritis patients. | Baseline
  To evaluate the frequency of LILRA3 in Ankylosing spondylitis and Axial psoriatic arthritis patients.

SECONDARY OUTCOMES:
Assosciation of LILRA3 with disease severity | Baseline
  To investigate the association of LILRA3 with Ankylosing spondylitis and Axial psoriatic arthritis disease activity and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Zahraa Abou eleyoun, PHD, Study Chair — Assiut University

REFERENCES:
- [Background] Ryu M, Chen Y, Qi J, Liu J, Fan Z, Nam G, Shi Y, Cheng H, Gao GF. LILRA3 binds both classical and non-classical HLA class I molecules but with reduced affinities compared to LILRB1/LILRB2: structural evidence. PLoS One. 2011 Apr 29;6(4):e19245. doi: 10.1371/journal.pone.0019245. PMID 21559424
- [Result] Wang R, Ward MM. Epidemiology of axial spondyloarthritis: an update. Curr Opin Rheumatol. 2018 Mar;30(2):137-143. doi: 10.1097/BOR.0000000000000475. PMID 29227352
- [Result] Poddubnyy D. Axial spondyloarthritis: is there a treatment of choice? Ther Adv Musculoskelet Dis. 2013 Feb;5(1):45-54. doi: 10.1177/1759720X12468658. PMID 23514983
- [Result] Norman PJ, Carey BS, Stephens HAF, Vaughan RW. DNA sequence variation and molecular genotyping of natural killer leukocyte immunoglobulin-like receptor, LILRA3. Immunogenetics. 2003 Jun;55(3):165-171. doi: 10.1007/s00251-003-0561-1. Epub 2003 May 16. PMID 12750859